CLINICAL TRIAL: NCT06555822
Title: A Phase I, Two-Part Study in Healthy Volunteers Consisting of a Randomized, Single-blind, Placebo-controlled Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of AZD5004 and a Randomized, Open-Label, Two-way Cross-over Study to Compare the Relative Bioavailability of Two Oral Tablet Strengths of AZD5004
Brief Title: A Study to Investigate Multiple Ascending Doses and Relative Bioavailability of AZD5004 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7260C00004
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants
Keywords: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Multiple Ascending dose (MAD) (AZD5004) (Experimental): Participants will receive repeated dosing of AZD5004 orally.
  Interventions: Drug: AZD5004
- Part A: Placebo (Placebo Comparator): Participants will receive matching Placebo orally.
  Interventions: Drug: Placebo
- Part B: Treatment 1 (AZD5004) (Experimental): Participants in Group 1 will receive Treatment 1 of AZD5004 and then Treatment 2 of AZD5004. Participants in Group 2 will receive Treatment 2 of AZD5004 and then Treatment 1 of AZD5004.
  Interventions: Drug: AZD5004
- Part B: Treatment 2 (AZD5004) (Experimental): Participants in Group 1 will receive Treatment 1 of AZD5004 and then Treatment 2 of AZD5004. Participants in Group 2 will receive Treatment 2 of AZD5004 and then Treatment 1 of AZD5004.
  Interventions: Drug: AZD5004

INTERVENTIONS:
Drug: AZD5004 — Participants will receive oral tablets of AZD5004 in Part A and Part B of the study as per arms they are assigned.
  Other Names: ECC5004
  Arms: Part A: Multiple Ascending dose (MAD) (AZD5004); Part B: Treatment 1 (AZD5004); Part B: Treatment 2 (AZD5004)
Drug: Placebo — Placebo will be administered as an oral tablet once daily.
  Arms: Part A: Placebo

SUMMARY:
The main purpose of this study is to assess the safety, tolerability, and pharmacokinetic (PK) of AZD5004 administered as multiple oral doses in healthy participants and to compare the relative bioavailability of two oral tablet strengths of AZD5004.

DETAILED DESCRIPTION:
This study comprises of 2 parts - Part A and Part B.

Part A is a placebo-controlled study to assess the safety, efficacy, tolerability, and PK of repeated dosing of AZD5004 compared with placebo.

Participants who are eligible according to the inclusion/exclusion criteria will be randomized to receive AZD5004 or matching placebo.

Part A will comprise:

1. A Screening Period of maximum 28 days.
2. A Treatment Period of 106 days.
3. A final Follow-up Visit approximately 14 days after the last study intervention administration.

Part B is a two-way cross-over study to compare the relative bioavailability of 2 oral tablet strengths of Formulation 1 (F1) of AZD5004.

The purpose of this study is to expand product knowledge between the 2 oral tablet strengths on plasma exposure levels to guide Phase 3 drug product development. The participants will be split into 2 groups. Group 1 will be dosed with Treatment 1 of AZD5004 and then dosed with Treatment 2 of AZD5004. Group 2 will be dosed with Treatment 2 of AZD5004 and then dosed with Treatment 1 of AZD5004.

Part B of the study will comprise:

1. A Screening Period of maximum 28 days.
2. Two Treatment Periods, each consisting of 7 days.
3. A final Follow-up Visit approximately 6 days after the last dose of study intervention administration.

ELIGIBILITY:
Inclusion Criteria:

* Must have suitable veins for cannulation or repeated venipuncture.
* Female(s) of Childbearing Potential must use adequate contraception (oral contraceptives are not permitted).
* Have a BMI ≥ 23 kg/m2 and not exceeding 35 kg/m2 inclusive and weigh at least 60 kg.
* No or off statin treatment for ≥ 4 weeks prior to the study treatment.

Exclusion Criteria:

* History of any clinically important disease or disorder.
* History of acute pancreatitis, chronic pancreatitis, gallstones, or elevation in serum lipase/pancreatic amylase.
* History or presence of gastrointestinal, hepatic, or renal disease.
* Clinically significant hepatic disease, inflammatory bowel disease, gastroparesis, severe disease, or surgery affecting the upper gastrointestinal tract.
* Any clinically important abnormalities in clinical chemistry, hematology, or urinalysis results.
* Any clinically important abnormalities in rhythm, blood pressure, heart rate, conduction or morphology of the resting electrocardiogram (ECG).
* Uncontrolled thyroid disease, defined as thyroid-stimulating hormone > 6.0 mIU/L or < 0.4 mIU/L at Screening.
* Current smokers or known history of alcohol or drug abuse.
* History of severe allergy/hypersensitivity or excessive intake of caffeine-containing drinks or food.
* Use of any prescribed or nonprescribed medication including antacids or analgesics.
* Participants who are on or are planning to undertake a weight loss program.
* History of psychosis, major depressive disorder, suicide attempt or suicidal ideation within the past year.
* Lactating, breastfeeding, or pregnant females or females who intend to become pregnant.
* Participants who are vegans or have medical dietary restrictions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Part A: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | From screening (Day -28) to last follow up visit (Day 120)
  To assess the safety and tolerability of AZD5004 following oral multiple ascending doses in healthy participants.
Part B: Maximum observed plasma (peak) drug concentration (Cmax) of AZD5004 | From Day 1 (Treatment Period 1) to Day 13 (end of Treatment Period 2)
  To evaluate the Cmax of 2 treatments of AZD5004 in healthy participants.
Part B: Area under the concentration-curve from time zero to the last quantifiable concentration (AUClast) | From Day 1 (Treatment Period 1) to Day 13 (end of Treatment Period 2)
  To evaluate the AUClast of 2 treatments of AZD5004 in healthy participants.
Part B: Area under concentration-time curve from time 0 to infinity (AUCinf) | From Day 1 (Treatment Period 1) to Day 13 (end of Treatment Period 2)
  To evaluate the AUCinf of 2 treatments of AZD5004 in healthy participants.
Part B: Time to reach maximum observed concentration (tmax) | From Day 1 (Treatment Period 1) to Day 13 (end of Treatment Period 2)
  To evaluate the tmax of 2 treatments of AZD5004 in healthy participants.

SECONDARY OUTCOMES:
Part A: Maximum observed plasma (peak) drug concentration (Cmax) of AZD5004 | From Day 1 to last follow up visit (Day 120)
  To characterize the Cmax of multiple ascending doses of AZD5004 in healthy participants.
Part A: Area under the concentration-curve from time zero to the last quantifiable concentration (AUClast) | From Day 1 to last follow up visit (Day 120)
  To characterize the AUClast of multiple ascending doses of AZD5004 in healthy participants.
Part A: Area under concentration time curve in the dosing interval (AUCtau) | From Day 1 to last follow up visit (Day 120)
  To characterize the AUCtau of multiple ascending doses of AZD5004 in healthy participants.
Part A: Amount of unchanged drug excreted into urine from time t1 to time t2 (Ae[t1-t2]) | From Day 1 to last follow up visit (Day 120)
  To characterize the Ae(t1-t2) of multiple ascending doses of AZD5004 in healthy participants.
Part A: Percentage of dose excreted unchanged in urine from time t1 to time t2 (fe[t1-t2]) | From Day 1 to last follow up visit (Day 120)
  To characterize the fe(t1-t2) of multiple ascending doses of AZD5004 in healthy participants.
Part A: Renal clearance (CLR) | From Day 1 to last follow up visit (Day 120)
  To characterize the CLR of multiple ascending doses of AZD5004 in healthy participants.
Part A: Percentage change from Baseline in body weight (kg) | Baseline (Day - 2) to Days 49, 91, and 106
  To assess the effects of AZD5004 compared to placebo on body weight change from baseline.
Part A: Absolute change from Baseline in body weight (kg) | Baseline (Day - 2) to Days 49, 91, and 106
  To assess the effects of AZD5004 compared to placebo on body weight change from baseline.
Part A: Percentage change from Baseline in Body Mass Index (BMI) (kg/m^2) | Baseline (Day - 2) to Days 49, 91, and 106
  To assess the effects of AZD5004 compared to placebo on body weight change from baseline.
Part A: Absolute change from Baseline in BMI (kg/m^2) | Baseline (Day - 2) to Days 49, 91, and 106
  To assess the effects of AZD5004 compared to placebo on body weight change from baseline.
Part B: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | From screening (Day -28) to last follow up visit (Day 14)
  To evaluate the safety and tolerability of 2 treatments of AZD5004 in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/